CLINICAL TRIAL: NCT03120260
Title: Comparing the Effect of Short Sleep Duration on Weight Loss of Overweight and Obese Women Attending a Weight Loss Program: A 12 Week Randomized Controlled Trial
Brief Title: Comparing Effect of Short Sleep Duration on Weight Loss of Overweight and Obese Women Attending a Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-201
Record Dates: First submitted 2017-04-15; First posted 2017-04-19 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Overweight
Keywords: Caloric Restriction; weight loss; sleep
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Sleep (Experimental): Diet+ have 5 hour sleep at night (SS)
  Interventions: Other: Diet
- Normal Sleep (Experimental): Diet+ have 7-8 hour sleep at night (NS)
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Intervention 'Diet+ short sleep versus normal sleep

SUMMARY:
The purpose of the present study is to evaluate the effect of sleep duration on weight loss of obese and overweight adult when they are in a weight loss plan (NovinDiet Protocol). The investigators aim is to compare the effects of short term sleep duration with normal sleep duration with respect to body weight (and abdominal adiposity).

ELIGIBILITY:
Inclusion Criteria:

* Must be female
* Must have < 7 hour sleep per night
* Must be 18-45 years of age.
* Must have Body mass index (BMI) between 27-35 kg/ m².
* Must be able to have moderate exercise.
* Must be interested to have weight loss.

Exclusion Criteria:

* Participating in a research project involving weight loss or physical activity in the previous six months.
* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medication that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 Weeks
  kg

SECONDARY OUTCOMES:
Body mass index reduction | 12 Weeks
  kg/m2
Fasting plasma glucose level | 12 Weeks
  mmol/l
lipid profiles | 12 Weeks
  mmol/l
Insulin resistance (HOMA) | 12 Weeks
  score
liver enzymes (SGOT, SGPT) | 12 Weeks
  U/l

CONTACTS AND LOCATIONS:
Locations (1):
- NovinDiet Clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided